CLINICAL TRIAL: NCT03664583
Title: ACHRU Community Partnership Program for Diabetes Self-Management for Older Adults - Canada
Acronym: ACHRU-CPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Maureen Markle-Reid, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: KPG 156883
Record Dates: First submitted 2018-08-23; First posted 2018-09-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Multiple Chronic Conditions; Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; Comorbidity; Aged; Health Services
MeSH Terms: conditions — Multiple Chronic Conditions; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A cross-jurisdictional, multi-site implementation-effectiveness type II hybrid randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomly assigned to the intervention group will be offered the ACHRU-Community Partnership Program (CPP) intervention in addition to usual primary care services offered by their local diabetes education centre or primary care setting. The CPP is a 6-month self-management intervention consisting of six core components: 1) home or virtual visits (up to 3) supported by phone calls by either a Registered Nurse (RN) or Registered Dietician (RD); 2) wellness sessions (up to 6, one per month) provided to patients and their caregivers at the location of the community partner or virtually; 3) monthly team case conferences with the provider team; 4) caregiver support; 5) collaboration with the primary care interprofessional team and other specialists; 6) nurse-led care coordination/system navigation.
  Interventions: Behavioral: ACHRU-Community Partnership Program (CPP)
- Control Group (No Intervention): Those who are randomly assigned to the control group will continue to be offered usual primary care services through their local diabetes education centre or primary care setting. The services that comprise usual diabetes care vary across the provinces e.g., length and focus of educational sessions, whether classes are strongly recommended versus optional (e.g., foot care, cardiac health, eating and exercise interventions), home visits, access to on-site professionals (e.g., endocrinologist, dietitian, physiotherapist, exercise specialist, pharmacist), connections with support services and community resources, and type of follow-up services available. Details of usual care provided at each site will be recorded.

INTERVENTIONS:
Behavioral: ACHRU-Community Partnership Program (CPP) — The intervention is a 6-month community navigation and self-management program for patients with diabetes and at least one additional chronic condition, and their caregivers, to improve health outcomes. The intervention will be provided by an interprofessional team of providers and consists of six core components.
  Arms: Intervention Group

SUMMARY:
Living with diabetes and other chronic (ongoing) conditions is common in older adults. These individuals have poorer health and higher use of health services compared to older adults with diabetes alone. Programs that help older adults self-manage their diabetes and other health conditions benefit both individuals and the healthcare system. The McMaster University Aging, Community and Health Research Unit developed and tested a new patient-centered, community-based program (CPP) to improve the delivery and outcomes of care for older adults with diabetes and other chronic conditions. This 6-month program was developed in partnership with patients, caregivers, primary and community care providers and researchers. The program is delivered by nurses, dietitians and community providers. It involves in-home or virtual visits by nurses and dietitians, monthly group wellness sessions at community centers or virtually, and monthly virtual team meetings. Wellness sessions include exercise, education, and social support. Caregivers are invited to be active participants along with patients. The program was successfully implemented in Ontario and Alberta. Participants who received the program had better quality of life, self-management, and mental health at no additional cost from a societal perspective compared to those receiving usual care. To determine how the program can best help people, more testing is needed with different communities and groups of people. We will partner with primary healthcare teams (e.g., family doctors' offices) in three provinces to adapt and test the program in a variety of real-world settings. We will assess how to best put this program into practice and measure outcomes important to patients and caregivers so study results are relevant to them. Study findings will guide the development of a plan for expanding the program to reach and benefit more older adults with diabetes and other chronic health conditions. Patients and caregivers will be involved as key partners in all aspects of the research.

DETAILED DESCRIPTION:
The purpose of this study is to examine the implementation and effectiveness of the CPP intervention in new settings and populations to demonstrate widespread effectiveness and ways to adapt CPP for diverse population subgroups and primary care setting and community care contexts. Based on the investigator's previous work, we expect that the CPP intervention will result in a greater improvement in mental health and will be cost neutral relative to usual care because program costs will be offset by lower use of other health services. A cross-jurisdictional, multi-site implementation-effectiveness type II hybrid randomized controlled trial will be conducted. The trial will be conducted in two sites in each of Ontario, Quebec, and Prince Edward Island. Each of the six sites will involve a primary care setting and a community care organization. Study participants will be randomly assigned to the intervention or usual care group. Participants randomly assigned to the intervention group will be offered the 6-month CPP intervention in addition to their usual primary care services offered by their local diabetes education centre or primary care setting. The primary outcome of intervention effectiveness is patient mental health. Other health outcomes for patients and their caregivers will be assessed (e.g., depression, anxiety, use of health and social services etc.). Implementation will be examined in-detail through qualitative evaluations with providers, patients and caregivers. Engagement of patients and caregivers will occur in all stages of the research study. Qualitative evaluation of patients and caregivers as research partners will be conducted through annual evaluations. Patient, Public (e.g., caregivers, knowledge users) and Community (e.g., local providers/representatives) Research Partners will be engaged in the research study by way of the study's established governance structures: Community Advisory Boards, Patient Advisory Council, and Steering Committee. Qualitative evaluation of Patient, Public and Community Research Partners will be conducted to inform implementation of the CPP intervention at the local context and the potential for widespread implementation and scale-up. Both quantitative and qualitative evaluations will be used to interpret study findings, and in the development of scale-up plans.

ELIGIBILITY:
Inclusion Criteria:

Patient participants ("CPP Target Population") will be included in the study if they meet the following inclusion criteria:

* Diagnosis of type 1 or type 2 diabetes
* Aged 65+ years
* Enrolled in a primary care organization
* Diagnosed with at least one other chronic condition
* Residing in the area served by the primary care and community site
* Capable of providing informed consent, or has a substitute decision-maker who is able to provide informed consent on his/her behalf
* Competent in English or has an interpreter who is competent in English for Ontario and Prince Edward Island (PEI) study sites. Patient participants that score 5 or higher on The Short Portable Mental Status Questionnaire (SPMSQ) will be eligible as patient participants. Those with scores below 5 will be eligible if they have a proxy decision-maker.

Caregiver participants will be included in the study if they meet the following inclusion criteria:

* Identified by the patient participant as an informal family or friend caregiver
* At least 18 years of age
* Provides physical, emotional, or financial care to the patient participant
* Scores 5 or higher on the SPMSQ

Provider and manager participants will be included in the study if they meet the following inclusion criteria:

* Working with the primary care setting or community partner organization at a study site
* Either a Registered Nurse (RNs) or Registered Dietitian (RDs) at the primary care setting
* A Program Coordinator (PC) from the community partner organization
* A manager of the RN or RD at the primary care setting
* A manager of the PC at the community partner organization

Patient, Public and Community Research Partner participants will be included in the study if they meet the following inclusion criteria:

* Older adult living in the community, or
* Community living family or friend caregiver of a person with a diagnosis of diabetes and one or more chronic condition, or
* Community living health provider or manager of persons with diabetes and one or more chronic condition, or
* A knowledge user (e.g. policy maker) who works in health planning or health policy decision making at the community level representative of study sites
* Persons not receiving the CPP intervention

Exclusion Criteria:

• Patient and caregiver participants in Ontario and PEI who do not speak English and do not have an interpreter/translator

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 295 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Mental Health Using the Short-Form 12 Health Survey Version 2 (SF-12v2) - Mental Component Summary score. | Baseline, 6-months
  The Short-Form 12 Health Survey Version 2 (SF-12v2) tool will be used to assess mental health. The tool consists of 12 questions that measure functional health and well-being from the participant's perspective. It provides scores for eight health domains (physical functioning, role-physical, bodily pain, general health, social functioning, role-emotional, mental health), by which a psychometrically-based Physical Component Summary (PCS) and Mental Component Summary (MCS) can be calculated. Response options include the frequency of feeling a certain way or behaviour across 3 or 5 categories (e.g., 'all of the time'...'none of the time'). Patients and caregivers will be evaluated for change in SF-12-MCS from baseline to 6-months. Total scale range: 0 - 100. Higher scores represent better mental functioning.

SECONDARY OUTCOMES:
Self-Management Using the Summary of Diabetes Self-Care Activities (SDSCA) | Baseline, 6-months
  The Summary of Diabetes Self-Care Activities (SDSCA) will be used to assess self-management. The SDSCA is a multidimensional measure of diabetes self-management with adequate internal and test-retest reliability, and evidence of validity and sensitivity to change. The revised SDSCA consists of 11 items that assess the following aspects of the diabetes regimen: (1) general and specific diet; (2) exercise; (3) blood-glucose testing; (4) foot care; and (5) smoking. Change in patient self-management will be evaluated using the SDSCA. Scale range: 0 - 71. Higher scores represent better self-management.
Physical Health Using the Short-Form 12 Health Survey Version 2 (SF-12v2) - Physical Component Summary score. | Baseline, 6-months
  The Short-Form 12 Health Survey Version 2 (SF-12v2) tool will be used to assess physical health. The tool consists of 12 questions that measure functional health and well-being from the participant's perspective. It provides scores for eight health domains (physical functioning, role-physical, bodily pain, general health, social functioning, role-emotional, mental health) by which a psychometrically-based Physical Component Summary (PCS) and Mental Component Summary (MCS) score can be calculated. Response options include the frequency of feeling a certain way or behaviour across 3 or 5 categories (e.g., 'all of the time'...'none of the time'). Patients and caregivers will be evaluated for change in SF-12-PCS from baseline to 6-months. Total scale range: 0 - 100. Higher scores represent better physical functioning.
Depressive Symptoms Using the Center for Epidemiologic Studies on Depression 10-Item Scale (CES-D-10) | Baseline, 6-months
  The Center for Epidemiologic Studies on Depression 10-Item Scale (CES-D-10) will be used to assess depressive symptoms. This tool has been used in prior studies of older adults with mood disorders, has a high degree of reliability and validity, and is a sensitive tool for measuring changes in depressive symptoms over time. Participants will be asked about the way they have felt or behaved in response to 10 statements such as 'I was happy'. Response options ask participants to select the frequency they have felt or behaved during the last week, ranging from 'rarely or none of the time (less than 1 day)', 'some or a little of the time (1-2 days)', 'occasionally or moderate (3-4 days)', to 'most or all of the time (5-7 days)'. Patients and caregivers will be evaluated for change in depressive symptoms using CES-D-10. Scale range: 0 - 30. Higher scores represent more depressive symptoms.
Level of Anxiety Using the Generalized Anxiety Disorder 7-Item (GAD-7) | Baseline, 6-months
  The Generalized Anxiety Disorder 7-Item (GAD-7) will be used to assess anxiety levels. The GAD-7 is a 7-item tool that asks about the type and frequency of being bothered by a list of problems. Response options include 'not at all', 'several days', 'more than half the days', or 'nearly every day', over the last two weeks. Patients and caregivers will be evaluated for change in level of anxiety using GAD-7. Scale range: 0 - 21. Higher scores represent more anxiety.
Physical Activity Using the Physical Activity Scale for the Elderly (PASE) | Baseline, 6-months
  The Physical Activity Scale for the Elderly (PASE) tool will be used to assess the physical activity of patients. The PASE measures physical activity over the past 7 days. It asks about the type and frequency of physical activity across categories of light, moderate and strenuous physical activity. Patients will be evaluated for change in physical activity using the PASE tool. Higher scores represent better physical activity.
Caregiver Strain Using the Modified Caregiver Strain Index (MCSI) | Baseline, 6-months
  The Modified Caregiver Strain Index (MCSI) will be used to assess caregiver strain. This tool will ask caregivers a list of 13 activities that they may have found to be difficult such as sleeping, physical strain, financial strain, personal plans, and work and family adjustments as a result of the caregiver role. Response options include 'yes' according to two levels, either 'yes, on a regular basis' or 'yes, sometimes', or alternatively, 'no'. Scale range: 0 - 26. Higher scores represent more strain.
Social Support Using the Abbreviated Duke Social Support Index (DSSI) | Baseline, 6-months
  The abbreviated, 11-item Duke Social Support Index (DSSI) will be used to measure social support. This 11-item instrument includes two major sub-scales: a 4-item social interaction sub-scale and a 7-item subjective support sub-scale. Response options on the social interaction sub-scale ask participants to rate the frequency of their social interactions in the past week: "none", "1-2", ">2", or "0-1 time", "2-5 times", "6 or more times". Response options on the subjective support sub-scale include "hardly ever", "some of the time", "most of the time", or "very dissatisfied", "somewhat dissatisfied" "satisfied". Scale range: 11-33. Higher DSSI scores represent more social support.
Functional Status Using the Duke Older Americans Resources and Services Procedures (OARS) Multidimensional Functional Assessment Questionnaire - Activities of Daily Living section | Baseline, 6-months
  The OARS Multidimensional Functional Assessment Questionnaire is a valid and reliable questionnaire, designed to assess the overall personal functional status and service use of older adults. Participants will be asked to respond to questions from the Activities of Daily Living section [14-items; activities of daily living (ADLs)/instrumental activities of daily living (IADLs)] of the OARS, which assesses both activities of daily living, such as eating, dressing and walking; and instrumental activities of daily living, such as using a telephone, shopping for groceries, and preparing meals. Response options include "without help", "with some help", and "completely unable". Scale range: 0-28. Higher scores represent a higher level of function.
Nutritional Status Using the Seniors in the Community Risk Evaluation for Eating and Nutrition tool (SCREEN II-AB) | Baseline, 6-months
  The Seniors in the Community Risk Evaluation for Eating and Nutrition tool (SCREEN II-AB) is an abbreviated, 8-item nutrition screening instrument for older adults living in the community, to identify individuals at risk for nutritional problems or who have poor nutritional status. Items assess for weight change in the past 6 months, intake of fruit, vegetables and fluid, meal consumption and preparation, appetite, and swallowing. Scale range: 0-52. Higher scores represent lower risk for nutritional problems.
Shared Decision-Making Using the CollaboRATE tool | Baseline, 6-months
  The CollaboRATE tool consists of 3 items that measure the level of shared decision-making in a clinical encounter from the patient's perspective. These items are: (i) How much effort was made to help you understand your health issues? (ii) How much effort was made to listen to what matters most to you about your health issues? (iii) How much effort was made to include what matters most to you in choosing what to do next? Participants are asked to rate their last appointment, on a 10-point scale from 0=No effort was made, to 9=Every effort was made. Scale range: 0-27. Higher scores represent a higher degree of shared decision-making.
Service Use Using the Health and Social Services Utilization Inventory (HSSUI) | Baseline, 6-months
  The Health and Social Services Utilization Inventory (HSSUI) will be used to assess service use of patients and caregivers. The HSSUI is a reliable and valid self-report questionnaire that measures the use of health and social services from a societal perspective. The HSSUI provides information on different categories of use including acute care service use such as emergency department visits and hospitalizations, use of nursing and allied health professionals, and visits to family doctors and specialists. As part of the HSSUI, diabetes and other medications, supplies and devices will also be assessed. Change in the use of health and social services will be assessed for patients and caregivers using the HSSUI. Patients (not caregivers) will be assessed for medication use using the HSSUI.
Glycated hemoglobin (HbA1c) | Baseline, 6-months
  Patients will be evaluated for glycated hemoglobin (HbA1c) as abstracted from their medical records. Values closest to the time frame will be used.
Glomerular Filtration Rate (GFR) | Baseline, 6-months
  Patients will be evaluated for glomerular filtration rate (GFR) as abstracted from their medical records. Values closest to the time frame will be used.
Low-Density Lipoprotein (LDL) | Baseline, 6-months
  Patients will be evaluated for low-density lipoprotein (LDL) as abstracted from their medical records. Values closest to the time frame will be used.
Collaboration Using the Partnership Self-Assessment Tool (PSAT) | 6-months
  The Partnership Self-Assessment (PSAT) will be used to assess the collaboration process. The PSAT tool has shown acceptable validity and reliability. Questions ask about different aspects of the partnership, and the strengths and weaknesses of the collaboration process involved in the partnership (e.g., synergy, leadership, efficiency, administration and management etc.). Providers and managers will be evaluated for change in collaboration. Scale range: 1 - 5. Lower scores represent a lower level of collaboration.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Markle-Reid, RN, PhD, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Scarborough Health Network, Scarborough Village, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University of Prince Edward Island, Charlottetown, Prince Edward Island
  - L'Universite Laval, Québec, Quebec

REFERENCES:
- [Derived] Fisher K, Carusone SC, Ganann R, Markle-Reid M, Northwood M, Sherifali D. Transforming healthcare by prioritizing qualitative and quantitative clinical trial evidence: evaluating the Aging, Community and Health Research Unit's Community Partnership Program for Older Adults (ACHRU-CPP). Trials. 2025 May 13;26(1):154. doi: 10.1186/s13063-025-08839-1. PMID 40361198
- [Derived] Northwood M, Chambers T, Fisher K, Ganann R, Markle-Reid M, Yous ML, Beleno R, Gaudet G, Gruneir A, Leung H, Lindsay C, Luebke K, Macartney G, Macatangay E, MacIntyre J, MacPhail C, Montelpare W, Morrison A, Shaffer L, St Pierre M, Tang F, Whiteside C. Readiness for scale up following effectiveness-implementation trial: results of scalability assessment of the Community Partnership Program for diabetes self-management for older adults with multiple chronic conditions. BMC Health Serv Res. 2025 Feb 20;25(1):284. doi: 10.1186/s12913-025-12378-5. PMID 39979911
- [Derived] Yous ML, Ganann R, Ploeg J, Markle-Reid M, Northwood M, Fisher K, Valaitis R, Chambers T, Montelpare W, Legare F, Beleno R, Gaudet G, Giacometti L, Levely D, Lindsay C, Morrison A, Tang F; ACHRU-CPP Research Team. Older adults' experiences and perceived impacts of the Aging, Community and Health Research Unit-Community Partnership Program (ACHRU-CPP) for diabetes self-management in Canada: a qualitative descriptive study. BMJ Open. 2023 Apr 5;13(4):e068694. doi: 10.1136/bmjopen-2022-068694. PMID 37019487
- [Derived] Ploeg J, Markle-Reid M, Valaitis R, Fisher K, Ganann R, Blais J, Chambers T, Connors R, Gruneir A, Legare F, MacIntyre J, Montelpare W, Paquette JS, Poitras ME, Riveroll A, Yous ML; ACHRU-CPP Research Team. The Aging, Community and Health Research Unit Community Partnership Program (ACHRU-CPP) for older adults with diabetes and multiple chronic conditions: study protocol for a randomized controlled trial. BMC Geriatr. 2022 Feb 4;22(1):99. doi: 10.1186/s12877-021-02651-7. PMID 35120457